CLINICAL TRIAL: NCT02949206
Title: A 3-Part First-in-Human Study to Assess the Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Pharmacodynamics of JNJ-64179375 in Healthy Male Subjects
Brief Title: A Study to Evaluate Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Pharmacodynamics of JNJ-64179375 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108238; 64179375EDI1001 (Other: Janssen Research & Development, LLC); 2016-003006-13 (EudraCT Number)
Record Dates: First submitted 2016-10-27; First posted 2016-10-31 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Part 1: Cohort 1 (0.03 mg/kg of JNJ-64179375 or Placebo) (Experimental): Participants in a ratio of 3:1 will receive a single 0.03 milligram per kilogram (mg/kg) intravenous (IV) dose of JNJ-64179375 or matching placebo on Day 1.
  Interventions: Drug: JNJ-64179375; Drug: Placebo
- Part 1: Cohort 2 (0.1 mg/kg of JNJ-64179375 or Placebo) (Experimental): Participants in a ratio of 3:1 will receive a single 0.1 mg/kg IV dose of JNJ-64179375 or matching placebo on Day 1.
  Interventions: Drug: JNJ-64179375; Drug: Placebo
- Part 1: Cohort 3 (0.3 mg/kg of JNJ-64179375 or Placebo) (Experimental): Participants in a ratio of 3:1 will receive a single 0.3 mg/kg IV dose of JNJ-64179375 or matching placebo on Day 1.
  Interventions: Drug: JNJ-64179375; Drug: Placebo
- Part 1: Cohort 4 (1.0 mg/kg of JNJ-64179375 or Placebo) (Experimental): Participants in a ratio of 3:1 will receive a single 1.0 mg/kg IV dose of JNJ-64179375 or matching placebo on Day 1.
  Interventions: Drug: JNJ-64179375; Drug: Placebo
- Part 1: Cohort 5 (2.5 mg/kg of JNJ-64179375 or Placebo) (Experimental): Participants in a ratio of 3:1 will receive a single 2.5 mg/kg IV dose of JNJ-64179375 or matching placebo on Day 1.
  Interventions: Drug: JNJ-64179375; Drug: Placebo
- Part 1: Cohort 6 (5.0 mg/kg of JNJ-64179375 or Placebo) (Experimental): Participants in a ratio of 3:1 will receive a single 5.0 mg/kg IV dose of JNJ-64179375 or matching placebo on Day 1.
  Interventions: Drug: JNJ-64179375; Drug: Placebo
- Part 1: Cohort 7 (Escalation Dose of JNJ-64179375 or Placebo) (Experimental): Dose escalation will proceed until the toxicology study exposure limits or a highest tolerable dose will be reached.
  Interventions: Drug: JNJ-64179375; Drug: Placebo
- Part 1: Cohort 8 (Escalation Dose of JNJ-64179375 or Placebo) (Experimental): Dose escalation will proceed until the toxicology study exposure limits or a highest tolerable dose will be reached.
  Interventions: Drug: JNJ-64179375; Drug: Placebo
- Part 2: Reversal Cohort :(50 IU/kg of 4-factor PCC) (Experimental): Participants will receive a 2.5 mg/kg of JNJ-64179375 or highest tolerable dose if lower than 2.5 mg/kg followed by administration of a single IV 50 International Unit per kilogram (IU/Kg) dose of a 4 factor prothrombin complex concentrate (PCC) or matching placebo on Day 1.
  Interventions: Drug: JNJ-64179375; Drug: Placebo; Drug: 4 Factor Prothrombin Complex Concentrate (PCC)
- Part 3: Subcutaneous Cohort (1.0 mg/kg of JNJ-64179375) (Experimental): Participants will receive a Single Subcutaneous (SC) dose of 1.0 mg.kg or highest tolerable dose if less than 1.0 mg/kg of JNJ-64179375 or matching placebo on Day 1.
  Interventions: Drug: JNJ-64179375; Drug: Placebo

INTERVENTIONS:
Drug: JNJ-64179375 — During part 1, participants will receive a single ascending Intravenous dose of JNJ-64179375 ranging from (0.03 mg/kg to 5.0 mg/kg). In Part 2, participants will receive a 2.5 mg/kg or highest tolerable dose if lower than 2.5 mg/kg of JNJ-64179375. In Part 3, participants will receive a Single Subcutaneous (SC) dose of 1.0 mg/kg or highest tolerable dose if less than 1.0 mg/kg of JNJ-64179375.
Drug: Placebo — Participants will randomly receive matching placebo in all 3 Parts on day 1 administered via IV Route (for Part 1 and 2) and SC route (for Part 3).
Drug: 4 Factor Prothrombin Complex Concentrate (PCC) — Following a single dose of JNJ-64179375, participants will receive a single IV dose of 4 factor-PCC.
  Arms: Part 2: Reversal Cohort :(50 IU/kg of 4-factor PCC)

SUMMARY:
The purpose of this study is to assess the safety and tolerability of JNJ-64179375 in Part 1 (Intravenous dose) and Part 3 (Subcutaneous dose) and potential for reversibility of JNJ-64179375 induced Pharmacodynamic effects on coagulation parameters and platelet function (Part 2) in healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index [weight kilogram per meter square (kg/m^2)] between 18 and 30 kg/m^2 (inclusive), and body weight greater than 50 kilogram (kg) but less than 100 kg
* Generally in good health on the basis of physical examination, medical history, vital signs, laboratory tests, and electrocardiogram (ECG) performed at screening and/or prior to administration of the initial dose of study drug
* Must sign an informed consent form (ICF) indicating that he understands the purpose of, and procedures required for, the study and is willing to participate in the study
* contraceptive use by men should be consistent with local regulations regarding the use of contraceptive methods for subject participating in clinical studies
* willing and able to adhere to the study visit schedule and other requirements, prohibitions, and restrictions specified in this protocol through the Day 113 visit

Exclusion Criteria:

* Acute illness, including an upper respiratory infection (with or without fever), within 7 days prior to study drug administration or have had a major illness or hospitalization within 1 month prior to study drug administration
* Clinically significant abnormal values for coagulation, hematology, clinical chemistry or urinalysis at screening or on Day -1 (at admission to the clinical research unit) as determined by the investigator or appropriate designee
* Have smoked tobacco or nicotine-related products within 6 months prior to dosing or does not agree to refrain through Day 113
* Donated blood or blood products or had substantial loss of blood [more than 500 milliliter (mL)] within 3 months before the first administration of study drug or intends to donate or donates blood or blood products during the study until 30 days after completion
* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, bleeding or thrombotic disorders

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2017-08-09 (Actual); Study Completion 2017-08-09 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of Participants With Adverse Events (AE) as a Measure of Safety and Tolerability | Up to Day 113
Part 3: Number of Participants With Adverse Events (AE) as a Measure of Safety and Tolerability | Up to Day 113
Part 2: Change From Baseline in Potential for Reversibility of the JNJ-64179375 Induced Pharmacodynamic Effects on Coagulation Parameters | Baseline and Day 1
  Change in Potential for Reversibility of the JNJ-64179375 will be assessed by assessing the change in thrombin time as coagulation parameter.
Part 2: Change From Baseline in Potential for Reversibility of the JNJ-64179375 Induced Pharmacodynamic Effects on Platelet Function | Baseline and Day 1
  Platelet function will be assessed by measuring platelet activation and aggregation in response to thrombin and other agonists and with the platelet function analyzer (PFA)100.

SECONDARY OUTCOMES:
Part 1 and 3: Maximum Observed Plasma Concentration (Cmax) of JNJ-64179375 | Predose, Day 1, 2, 4, 7, 10, 14, 22, 29, 43, 57, 85 and 113
  Cmax is defined as maximum observed plasma concentration of JNJ-64179375.
Part 1 and 3: Area Under the Plasma Concentration-Time Curve From Time Zero to Time of the Last Quantifiable Concentration (AUClast) of JNJ-64179375 | Predose, Day 1, 2, 4, 7, 10, 14, 22, 29, 43, 57, 85 and 113
  The (AUC [0-last]) is defined as Area under the plasma concentration versus time curve from time 0 to the time corresponding to the last quantifiable serum concentration of JNJ-64179375.
Part 1 and 3: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of JNJ-64179375 | Predose, Day 1, 2, 4, 7, 10, 14, 22, 29, 43, 57, 85 and 113
  The (AUC [0-infinity]) is defined as Area under the plasma concentration versus time curve from time 0 to infinity with extrapolation of the terminal phase.
Part 1 and 3: Terminal Half-Life (t1/2) of JNJ-64179375 | Predose, Day 1, 2, 4, 7, 10, 14, 22, 29, 43, 57, 85 and 113
  Half-life (t[1/2]) is associated with the terminal slope (lambda [z]) of the semi-logarithmic drug concentration-time curve, calculated as 0.693/lambda(z).
Part 1: Total Systemic Clearance (CL) of JNJ-64179375 | Predose, Day 1, 2, 4, 7, 10, 14, 22, 29, 43, 57, 85 and 113
  CL is defined as total systemic clearance after intravenous administration of JNJ-64179375.
Part 1: Apparent Volume of Distribution at Terminal Phase After Intravenous Administration (Vz) of JNJ-64179375 | Predose, Day 1, 2, 4, 7, 10, 14, 22, 29, 43, 57, 85 and 113
  Vz is defined as the Apparent volume of distribution at terminal phase after intravenous administration.
Part 3: Time to Reach Maximum Observed Concentration (Tmax) of JNJ-64179375 | Predose, Day 1, 2, 4, 7, 10, 14, 22, 29, 43, 57, 85 and 113
  Tmax is defined as time to the maximum observed plasma concentration of JNJ-64179375.
Part 3: Total Systemic Clearance Over Bioavailability After Subcutaneous (SC) Administration (CL/F) of JNJ-64179375 | Predose, Day 1, 2, 4, 7, 10, 14, 22, 29, 43, 57, 85 and 113
  CL/F is defined as total systemic clearance over bioavailability after SC administration.
Part 3: Apparent Volume of Distribution at Terminal Phase Over Bioavailability After Subcutaneous Administration (Vz/F) of JNJ-64179375 | Predose, Day 1, 2, 4, 7, 10, 14, 22, 29, 43, 57, 85 and 113
  (Vz/F) is defined as Apparent Volume of distribution at terminal phase over bioavailability after SC administration of JNJ-64179375.
Part 3: Absolute Bioavailability (F) After Subcutaneous Administration of JNJ-64179375 | Predose, Day 1, 2, 4, 7, 10, 14, 22, 29, 43, 57, 85 and 113
  F is defined as absolute bioavailability after SC administration of JNJ-64179375.
Part 1 and 3: Immunogenicity of JNJ-64179375 | Predose, Day 7, 14, 29, 57, 85 and 113
  Plasma samples will be collected and screened for antibodies binding to JNJ-64179375 and the titer of confirmed positive samples will be reported.
Part 2: Maximum Observed Plasma Concentration (Cmax) of JNJ-64179375 in presence of 4-factor prothrombin complex concentrate (PCC) | Predose, Day 1, 2, 4, 7, 10, 14, 22, 29, 43, 57, 85 and 113
  Cmax is defined as maximum observed plasma concentration of JNJ-64179375.
Part 2: Area Under the Plasma ConcentrationTime Curve From Time Zero to Time of the Last Quantifiable Concentration (AUC [0-last]) of JNJ-64179375 in the presence of 4-factor PCC | Predose, Day 1, 2, 4, 7, 10, 14, 22, 29, 43, 57, 85 and 113
  The (AUC [0-last]) is defined as Area under the plasma concentration versus time curve from time 0 to the time corresponding to the last quantifiable serum concentration of JNJ-64179375
Part 2: Area Under the Plasma ConcentrationTime Curve From Time Zero to Infinite Time (AUC [0-infinity]) of JNJ-64179375 in the presence of 4-factor PCC | Predose, Day 1, 2, 4, 7, 10, 14, 22, 29, 43, 57, 85 and 113
  The (AUC [0-infinity]) is defined as Area under the plasma concentration versus time curve from time 0 to infinity with extrapolation of the terminal phase.
Part 2: Terminal Half Life [t(1/2)] of JNJ-64179375 in the presence of 4-factor PCC | Predose, Day 1, 2, 4, 7, 10, 14, 22, 29, 43, 57, 85 and 113
  Half life [t(1/2)] is associated with the terminal slope (lambda [z]) of the semilogarithmic drug concentration time curve, calculated as 0.693/lambda(z).
Part 2: Total Systemic Clearance (CL) of JNJ-64179375 in the presence of 4-factor PCC | Predose, Day 1, 2, 4, 7, 10, 14, 22, 29, 43, 57, 85 and 113
  CL is defined as total systemic clearance after intravenous administration of JNJ-64179375.
Part 2: Apparent Volume of Distribution at Terminal Phase After Intravenous Administration (Vz) of JNJ-64179375 in the presence of 4-factor PCC | Predose, Day 1, 2, 4, 7, 10, 14, 22, 29, 43, 57, 85 and 113
  Vz is defined as the Apparent volume of distribution at terminal phase after intravenous administration.
Part 2: Immunogenicity of JNJ-64179375 in the presence of 4-factor PCC | Predose, Day 7, 14, 29, 57, 85 and 113
  Plasma samples will be collected and screened for antibodies binding to JNJ-64179375 and the titer of confirmed positive samples will be reported.
Part 2: Number of Participants With Adverse Events (AE) as a Measure of Safety and Tolerability | Baseline to End of treatment (Day 113)
Part 1 and 3: Pharmacodynamic Effect of JNJ-64179375 on Platelet Function | Predose, Day 1, 2, 4, 7, 14, 29, 57 and 113
  Platelet function will be assessed by measuring platelet activation and aggregation in response to thrombin and other agonists and with the platelet function analyzer (PFA)-100.
Part 1 and 3: Pharmacodynamic Effect of JNJ-64179375 on Coagulation Parameters | Predose, Day 1, 2, 4, 7, 14, 29, 57 and 113
  The pharmacodynamic effect of JNJ-64179375 on coagulation parameters will be assessed by measuring the change in thrombin time.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium